CLINICAL TRIAL: NCT03690908
Title: Infraorbital Nerve Involvement on Magnetic Resonance Imaging in European Patients With IgG4-related Ophthalmic Disease
Brief Title: Infraorbital Nerve Involvement on Magnetic Resonance Imaging in IgG4-related Ophthalmic Disease
Acronym: RetroG4
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NI_2016_1_ALR
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: IgG4-related Disease; Orbital Infections, Inflammations and Irritations
MeSH Terms: conditions — Immunoglobulin G4-Related Disease; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IgG4-related orbital inflammation: patients with orbital inflammation and positive IgG4 immunostaining in orbital biopsy
  Interventions: Other: no intervention (descriptive study)
- non IgG4-related orbital inflammation: patients with orbital inflammation and negative IgG4 immunostaining in orbital biopsy
  Interventions: Other: no intervention (descriptive study)

INTERVENTIONS:
Other: no intervention (descriptive study) — no intervention (descriptive study)

SUMMARY:
Infraorbital nerve enlargement (IONE) on magnetic resonance imaging is known to be a possible consequence of IgG4-related ophthalmic disease. However this imaging sign can also be found in other conditions causing orbital inflammation. This study aims at comparing the frequency of IONE in patients suffering from IgG4-related ophthalmic disease (IgG4-ROD) versus patients suffering from non-IgG4-related ophthalmic disease (non-IgG4-ROD)

ELIGIBILITY:
Inclusion criteria :

* Patient aged 18 and older treated in Fondation Rothschild (tertiary ophthalmology facility, Paris, France) from January 2006 through April 2015
* Presence of a clinical orbital inflammation: mass/swelling, pain, exophthalmos, visual loss, ptosis, or diplopia.
* The presence of at least one pretherapeutic MRI confirming the inflammation of one or more orbital structures: the lacrimal gland, fat, muscles, or infraorbital nerve. The mandatory minimal MRI protocol include the following sequences: T1- and T2-weighted MRI image, in the transverse and coronal plane, and a fat-suppressed T1-weighted image in the coronal plane obtained after intravenous administration of a gadolinium chelate.
* Completion of at least one orbital biopsy with a pathologic examination and an immunohistochemical screen for IgG4.

Exclusion criteria :

* Clinical and biological signs of thyroid-associated orbitopathy
* Histologically proven lymphoma
* Pretherapeutic MRI that is insufficient for an adequate interpretation
* Absence of IgG4 testing in the pathology examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients suffering from non-thyroid, non-lymphoma related orbital inflammation treated in Fondation Rothschild (tertiary ophtalmology facility, Paris, France) from January 2006 through April 2015.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with infraorbital nerve involvement in magnetic resonance imaging | Within 2 weeks after the first consultation for orbital inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rotchschild, Paris, France

IPD SHARING:
Plan to Share IPD: No